CLINICAL TRIAL: NCT01187927
Title: Drug Use Investigation for Cervarix®
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114332
Record Dates: First submitted 2010-08-20; First posted 2010-08-24 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Infections, Papillomavirus
MeSH Terms: conditions — Papillomavirus Infections | interventions — human papillomavirus vaccine, L1 type 16, 18

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Female subjects: Subjects received Cervarix® as per routine practice
  Interventions: Biological: Cervarix®

INTERVENTIONS:
Biological: Cervarix® — Administered according to the prescribing information in the locally approved label by the authorities.

SUMMARY:
This post-marketing study was designed to assess safety and efficacy of Cervarix® vaccine in Japanese female subjects under conditions of actual use.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be female
* Subject must be aged 10 and over

Exclusion Criteria:

* Subject with obvious fever
* Subject with obvious severe acute disease
* Subject with hypersensitivity to any component of Cervarix®
* Other than above, subject who is in inappropriate conditions for vaccination

Min Age: 10 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Japanese women who received Cervarix® for the first time
Sampling Method: Probability Sample
Enrollment: 1230 (Actual)
Dates: Start 2010-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
The number of subjects with solicited local adverse events | 7 days after vaccination
  Local adverse events: pain, redness, swelling at the vaccination site
The number of subjects with solicited general adverse events | 7 days after vaccination
  General adverse events: fatigue, fever, gastrointestinal symptoms (nausea, vomiting, diarrhea, abdominal pain, etc.), headache, arthralgia, myalgia, urticaria, and rash
The number of subjects with unsolicited adverse events | 30 days after vaccination
  Any symptoms other than specified (local/systemic) symptoms
The number of subjects with serious adverse events | 30 days after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline